CLINICAL TRIAL: NCT03174457
Title: Non-interventional Study on the Safety and Efficacy for Prevention and Treatment of Fungal Infections in Paediatric Patients in Asia/Oceania - ERADICATE Study
Brief Title: Non-interventional Study for Prevention and Treatment of Fungal Infections in Paediatric Patients in Asia/Oceania - ERADICATE Study
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Singapore Pte. Ltd. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: 9463-MA-1006
Record Dates: First submitted 2017-05-31; First posted 2017-06-02 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2018-10

CONDITIONS: Invasive Fungal Infections
Keywords: Oesophageal Candidiasis; Paediatric; Invasive Candidiasis; Prophylaxis of Candida Infections; Candidemia; Aspergillosis; Micafungin
MeSH Terms: conditions — Invasive Fungal Infections; Candidiasis, Invasive; Candidemia; Aspergillosis | interventions — Micafungin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Treatment: micafungin: Participants receive once daily by intravenous infusion.
  Interventions: Drug: Micafungin

INTERVENTIONS:
Drug: Micafungin — Intravenous
  Other Names: micafungin sodium; Mycamine; FK463

SUMMARY:
The aim of the study is to prospectively evaluate the safety and efficacy of micafungin when prescribed for prophylaxis or treatment of fungal infections in different real-world clinical conditions and centers, in pediatric patients in Asia/Oceania.

DETAILED DESCRIPTION:
The study will collect safety and efficacy data from pediatric patients who are prescribed intravenous micafungin for prophylaxis. During this trial, patients with two separate indications will be treated. The first, Invasive candidiasis will have a minimum treatment of 2 weeks. The second, Oesophageal candidiasis will have a minimum treatment of 1 week. Both indications will have a follow-up period of 4 weeks after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Prescribed micafungin for prophylaxis or treatment of fungal infections.

According to treatment guidelines, micafungin may not be a suitable treatment for the following patients:

* The patient has evidence of impaired liver function: alanine aminotransferase (AST), aspartate aminotransferase (ALT) >5 times the upper limit of normal (ULN) or total bilirubin >2 times ULN.
* The patient has a history of allergy, hypersensitivity, or any serious reaction to the echinocandin class of antifungals.
* The patient has a confirmed systemic fungal infection with a non-Candida species.

Exclusion Criteria:

* The patient is receiving micafungin treatment in combination with other antifungal drugs.

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Paediatric patients for whom micafungin is prescribed for prophylaxis or treatment of fungal infections
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2017-06-21 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of Adverse Drug Reactions (ADRs) collected during the observational period | Up to end of trial (up to 95 weeks)
  ADR is considered to be any noxious and unintended response associated with the use of a drug in humans, at any dose, where a causal relationship (drug-event) is at least a reasonable possibility
Safety assessed by incidence of Serious Adverse Events (SAEs) | Up to end of trial (up to 95 weeks)
  Adverse event (AE) is considered "serious" if the investigator or sponsor view any of the following outcomes: Death, life-threatening, persistent or significant disability/incapacity, congenital anomaly or birth defect, hospitalization, or medically important event
Incidence of death attributable to micafungin treatment | Up to end of trial (up to 95 weeks)
  Death, if considered by the clinician to be attributable to micafungin
Safety assessed by vital sign measurements | Up to end of trial (up to 95 weeks)
  Vital sign measurements include systolic and diastolic blood pressure, pulse rate, and body temperature
Safety assessed by AEs of special interest (stratified by relationship to micafungin treatment) | Up to end of trial (up to 95 weeks)
  This includes hepatic dysfunction, renal dysfunction, infusion-related reactions, haemolytic events, histamine-release/allergic-type reactions and injection site reactions

SECONDARY OUTCOMES:
Safety assessed by nature, frequency and severity of Adverse Events (AEs) | Up to end of trial (up to 95 weeks)
  Adverse events (AEs) will be coded using the Medical Dictionary for Regulatory Activities (MedDRA). AEs that started or worsened during the observational period after the start of micafungin treatment will be summarized by the time period of onset. AE occurring within 3 days after end of therapy will be defined as treatment emergent adverse events
Overall treatment success | Up to end of trial (up to 95 weeks)
  The overall treatment success will be defined as a complete or partial clinical response in proven fungal infection, and by an empirical treatment composite outcome score in probable/possible fungal infection. Overall treatment success for patients receiving prophylactic treatment is defined as the absence of proven, probable, possible or suspected Invasive Fungal Infection (IFI) during the period of prophylactic therapy and up to 4 weeks after stopping micafungin administration
Change from baseline to end of treatment in safety laboratory parameters | Up to end of trial (up to 95 weeks)
  Indication of hepatic or renal dysfunction
Mycological response at end of treatment in patients with proven invasive fungal infection with candida or aspergillus species | Up to end of trial (up to 95 weeks)
  Response will be defined as eradication, presumed eradication, or overall

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Singapore Pte. Ltd.
Locations (16):
- Hong Kong (2):
  - Site HK203, New Territories
  - Site HK202, Pok Fu Lam
- Site SG801, Singapore, Singapore
- South Korea (4):
  - Site KR401, Seoul
  - Site KR402, Seoul
  - Site KR403, Seoul
  - Site KR404, Seoul
- Taiwan (6):
  - Site TW606, Changhua
  - Site TW603, Taichung
  - Site TW605, Taichung
  - Site TW601, Taipei
  - Site TW604, Taipei
  - Site TW602, Taoyuan District
- Thailand (3):
  - Site TH701, Bangkok
  - Site TH703, Bangkok
  - Site TH704, Chiang Mai

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.